CLINICAL TRIAL: NCT04291365
Title: Assessing the Use of Alternative Methods of Blood Pressure Measurement in Obstetric Patients
Brief Title: Alternative Blood Pressure Measurements in OB Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Tara Lynch, Assistant Professor, Albany Medical College
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5736
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Obesity; Blood Pressure
MeSH Terms: conditions — Obesity | interventions — Blood Pressure Determination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normal weight (Other)
  Interventions: Diagnostic Test: Blood pressure measurement
- Obesity Class 1 (Other)
  Interventions: Diagnostic Test: Blood pressure measurement
- Obesity Class 2 (Other)
  Interventions: Diagnostic Test: Blood pressure measurement
- Obesity Class 3 (Other)
  Interventions: Diagnostic Test: Blood pressure measurement

INTERVENTIONS:
Diagnostic Test: Blood pressure measurement — Study subjects will have a total of 9 blood pressure measurements taken (3 on upper arm, 3 on lower arm, and 3 on wrist)

SUMMARY:
The incidence of obesity has been increasing worldwide. In women with obesity, the anthropometric differences in the distribution of subcutaneous tissue can make accurate measurement of blood pressure difficult. A large upper arm circumference can prevent the use of a brachial artery blood pressure cuff and often prompts the use of alternative methods for blood pressure measurement, including measurements on the wrist or forearm. Outside of the obstetric population, there is evidence that if measurement of the blood pressure at the upper arm is not possible then measurement at the wrist can be used. Despite this evidence in non-pregnant patients, there is limited evidence in pregnancy regarding the accuracy of blood pressure measurements on the forearm or wrist. Accurate measurement of blood pressure is especially important in pregnancy to allow for prompt treatment of severe hypertension and for accurate diagnosis of hypertensive disorders of pregnancy. Error in measurement could lead to iatrogenic preterm birth or under treatment of severe hypertension, both which can lead to severe maternal and fetal morbidity and mortality. Additionally, it is biologically plausible that an increase in subcutaneous edema and vascular changes in pregnancy could lead to a larger discrepancy in blood pressure measurements between upper arm, forearm and wrist measurements.

Due to the increasing epidemic of obesity and the increasing need for accurate alternative blood pressure measurements the investigators propose a prospective observational study of pregnant women ≥18 years old admitted to labor and delivery for any indication or seen for prenatal care in OBGYN clinic. A total of 20 women in each BMI class (normal, overweight (25-29.9), class 1 (30-34.9), class 2 (35-39.9), class 3 (>40) will be enrolled (100 total). Participation will include a total of 9 blood pressure measurements, biometric measurements on the patient's upper arm, forearm, and wrist and a brief questionnaire. The investigators hypothesize that there will be a discrepancy between blood pressure measurements on the upper arm and forearm or wrist.

ELIGIBILITY:
Inclusion Criteria:

* >=18 years old
* prenatal care at study hospital
* english speaking

Exclusion Criteria:

* Age <18
* Active upper extremity DVT
* Inability to measure blood pressure on arm
* Unable to give consent

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure brachial | 1 day
Blood pressure radial | 1 day
Blood pressure wrist | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Tara Lynch, MD, Principal Investigator — Albany Medical College
Locations (1):
- Albany Medical Center, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lende MN, Feustel PJ, Alafifi RL, Lynch TA. Impact of obesity on blood pressures measured at alternative locations during pregnancy. Am J Obstet Gynecol MFM. 2021 Sep;3(5):100441. doi: 10.1016/j.ajogmf.2021.100441. Epub 2021 Jul 3. PMID 34229125